CLINICAL TRIAL: NCT07141628
Title: Etude de l'hyperlipoprotéinémie A Comme Marqueur de Risque Cardio-vasculaire Chez Les Patients Atteints de Maladie rénale Chronique au Stade 4
Brief Title: Hyperlipoproteinemia A as a Marker of Cardiovascular Risk in Patients With Stage 4 Chronic Kidney Disease
Acronym: LPACKD45
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2024-2/OM01
Record Dates: First submitted 2025-08-19; First posted 2025-08-26 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-08

CONDITIONS: CKD; Cardiovascular Diseases
Keywords: lipoproteinA
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stage 4 chronic kidney disease without replacement therapy
  Interventions: Diagnostic Test: lipoprotein A level dosing

INTERVENTIONS:
Diagnostic Test: lipoprotein A level dosing — Plasma levels measured in mmol/l

SUMMARY:
The blood level of lipoprotein A (Lp(a)) is linked to mutations in gene 6 and is associated with atherothrombotic risk and clinical manifestations such as myocardial infarction, ischemic stroke, and aortic valve calcification and stenosis. Several studies show an increased cardiovascular risk for a level >125 nmol/L. Patients with severe chronic kidney disease (CKD) or on hemodialysis are at high cardiovascular risk, and Lp(a) levels would allow for better reclassification of this cardiovascular risk in the general population.

The study authors wished to the heterogeneity of the Lp(a) level in the population with CKD stages 4 without renal replacement therapy and to identify whether a high Lp(a) level is associated with cardiovascular comorbidity defined by the presence of cardiovascular comorbidity after adjustment for known risk factors such as diabetic status, obesity, smoking, LDLc level and medical treatment for cardiovascular prevention (statins, etc.). Furthermore, they will evaluate whether there is a link between a high level (> 125 mmol/l) of Lp(a) at inclusion in the cohort and the occurrence of cardiovascular or renal events (i.e. death of cardiovascular origin or occurrence of MI, stroke, stage 4 peripheral artery disease (PAD) or initiation of renal replacement) over a follow-up period of 18 months which could raise questions about the benefit of a specific treatment which remains to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Patient being followed at the Nîmes University Hospital for stage 4 chronic kidney disease without replacement therapy
* Patient available for follow-up at 18 months

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Familial hypercholesterolemia
* Morbid obesity (BMI > 40 kg/m2).
* Persons deprived of their liberty by a judicial or administrative decision, persons receiving psychiatric care, and persons admitted to a health or social care facility for purposes other than research (Article L1121-6 of the French Public Health Code)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage 4 chronic kidney disease without replacement therapy followed as outpatients at Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Link between hyperlipoproteinemia A and a first event of cardiovascular death | 18 months
  cardiovascular death: yes/no
Link between hyperlipoproteinemia A and a first event of myocardial infarction | 18 months
  myocardial infarction: yes/no
Link between hyperlipoproteinemia A and a first event of stroke | 18 months
  stroke: yes/no
Link between hyperlipoproteinemia A and a first event of peripheral artery disease stage 4 | 18 months
  peripheral artery disease stage 4: yes/no
Link between hyperlipoproteinemia A and a first event of initiation of renal replacement therapy | 18 months
  initiation of renal replacement therapy: yes/no

SECONDARY OUTCOMES:
Rate of hyperlipoproteinemia A | Baseline (Day 0)
  defined as a lipoprotein A level > 125 nmol/L
Link between hyperlipoproteinemia A and a history of ischemic heart disease at inclusion | Baseline (Day 0)
  Ischemic heart disease: yes/no
Link between hyperlipoproteinemia A and a history ischemic stroke at inclusion | Baseline (Day 0)
  Ischemic stroke: yes/no
Link between hyperlipoproteinemia A and a history of calcified aortic stenosis at includion | Baseline (Day 0)
  Calcified aortic stenosis: yes/no
Link between hyperlipoproteinemia A and a history of lower limb arterial disease stage 2-4 at inclusion | Baseline (Day 0)
  Lower limb arterial disease stage 2-4: yes/no
Link between hyperlipoproteinemia A and a history of vascular nephropathy at inclusion | Baseline (Day 0)
  Vascular nephropathy: yes/no
Link between hyperlipoproteinemia A and a history of arterial angioplasty at any site at inclusion | Month 18
  coronary artery or limb angioplasty: yes/no
Link between hyperlipoproteinemia A and hospitalization for cardiac decompensation during follow-up | Month 18
  hospitalization for cardiac decompensation: yes/no
Link between hyperlipoproteinemia A and the occurrence of repeated cardiovascular events during follow-up | Month 18
  Cumulative events from the following: myocardial infarction, stroke, PAD stage 4, initiation of renal replacement therapy, death, arterial angioplasty at any site, cardiac decompensation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Moranne, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France